CLINICAL TRIAL: NCT05721352
Title: Arthritis Pain Reduction in Older Adults
Brief Title: Arthritis Ease Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Linda Larkey, Professor, Arizona State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00013939
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis; Chronic Pain; Kinesiophobia
Keywords: Heart Rate Variability; Biofeedback; Virtual Reality; Body awareness; Self regulation
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Kinesiophobia; Self-Control

STUDY DESIGN:
Intervention Model Description: Single-group pre-post intervention design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): * All participants will receive access to the phone application with a virtual reality headset and heart rate variability Bluetooth ear sensor.
  * Participants will be instructed to download a free phone app Elite Heart Rate Variability, login using study provided de-identified research email address, pair the Bluetooth ear sensor and record a five-minute resting heart rate variability reading at baseline and each time point of the study prior to beginning intervention.
  * Participants will be asked to use the intervention phone application for 7-10 minute sessions twice daily 5 days a week for 8 weeks.
  * For the first 8 weeks, participants will receive brief, daily texts encouraging participation in the smart phone application.
  * During weeks 9 through 12, will receive relaxation reminders daily via text to determine if use is sustained past the intervention phase
  Interventions: Behavioral: Virtual Reality Nature scene plus heart rate variability biofeedback phone application

INTERVENTIONS:
Behavioral: Virtual Reality Nature scene plus heart rate variability biofeedback phone application — phone app for slow- paced breath training with biofeedback in a virtual reality nature scene

SUMMARY:
The goal of this clinical trial is to test using a pain and anxiety reduction phone application in older adults with knee osteoarthritis and chronic pain. The main questions it seeks to answer are:

1. How acceptable is using a phone app in older adults with knee osteoarthritis and chronic pain to lower pain, pain stress and reduce fear of movement?
2. What are the effects of combining biofeedback with a virtual reality nature scene and paced breath training to increase heart rate variability on pain and anxiety among older adults with knee osteoarthritis?
3. What is the role of self-regulation and body awareness in predicting or strengthening the effect of combining virtual reality, heart rate variability biofeedback in older adults with knee osteoarthritis?.

Participants will be asked to:

1. use a phone application for 7-10 minute sessions twice daily 5 days a week for 8 weeks.
2. receive relaxation reminders weeks 9 through 12 to see if use continues past the intervention phase.
3. complete surveys describing pain, physical activity, fear of movement, body awareness and self-regulation, pain stress pre/post the app use.
4. complete a survey and interview after 8 weeks of phone app use to describe the experience of its use.

DETAILED DESCRIPTION:
Purpose: This single-group pre-post intervention design, study will explore the feasibility of using a multicomponent phone-based app for 8 weeks to reduce pain, pain stress effects, decreased heart rate variability and fear of movement in 24 older adults with knee osteoarthritis and to examine sustained use and or effects at 4 weeks after intervention period.

Aim 1 Evaluate the feasibility (adherence and satisfaction) of a multicomponent phone app combining virtual reality and heart rate variability biofeedback for use in older adults with knee osteoarthritis and chronic pain and gain descriptive evaluations of the experience in exit interviews.

Adherence: The adherence benchmark will be 80% of participants will participate at least 5 days per week during the initial 8-week intervention period. Adherence will be examined (not benchmarked) during the 4-week follow-up period.

Satisfaction: Exit interviews will demonstrate that 80% of participants practicing with the phone app rate the experience as satisfying or highly satisfying.

Aim 2 Evaluate the preliminary effects of multicomponent phone app use (5 days a week for 8 weeks) in older adults with knee osteoarthritis, in relation to pain, pain stress effects, and fear of movement (kinesiophobia), and examine sustained use patterns and effects with only reminders from the app during the 4-week follow-up period.

Aim 3: Examine the role of body awareness and self-regulation to moderate (predict) or mediate (strengthen) the effect of a virtual reality nature scene and heart rate variability biofeedback phone application in older adults with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults
* Diagnosed osteoarthritis of the knee(s)
* smart phone access
* Pain scale rating of 4-10 on the numerical pain rating scale (0- 10) \
* Pain duration of 3 months or greater
* Score of 15 or greater on the Tampa Scale of Kinesiophobia (fear of movement) scale

Eligibility includes:

* Willingness to engage in the study for 8 weeks
* Being available for 1-3 phone calls for data collection at pre- and post-8-week intervention and at 4 weeks post-intervention conclusion

Exclusion criteria:

* Self-report of: acute illness,
* Cancer
* HIV
* Systemic inflammatory disease (rheumatoid arthritis, lupus)
* History of neurologic disease, seizure disorder,
* Current or history of mental illness illness with hallucinations
* Motion sickness or vestibular disorders
* Acute or chronic respiratory disease
* Dysrhythmic heart disease
* Beta or calcium channel blocker medication use
* Monovision \\
* Current use of Heart rate variability training activities will also be excluded

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Adherence Measure | 8 weeks
  The adherence benchmark will be 80% of participants will participate at least 5 days per week during the initial 8-week intervention period. Adherence will be examined (not benchmarked) during the 4-week follow-up period
Satisfaction Measure | 8-12 Weeks
  Exit interviews will demonstrate that 80% of participants practicing with the phone app rate the experience as satisfying or highly satisfying

SECONDARY OUTCOMES:
Patient-reported outcomes measurement information -29 v2.0 system-29 Profile v2.0 | Baseline, 4, 8 and 12 weeks
  The Patient-reported outcomes measurement information -29 v2.0 profile assesses pain intensity using a single 0-10 numeric rating item (lower score is better) and seven physical and mental health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. Each question has a 5 point Likert scale and each domain has a minimum score of 4 and a maximum score of 20,,with higher score being better.is no composite score as individual items are scored within each health domain.
Multidimensional Assessment of Somatic Sense Scale | Baseline, 4, 8 and 12 weeks
  8 Scale (32 items) Self-report measure of dimensions of body awareness and self regulation (noticing, not distracting, not worrying, attention regulation, attention regulation, emotional awareness, body listening, trust and self regulation) Each scale has a 0-5 point Likert Scale with higher numbers being better. The range for each scale score mean is derived and compared to baseline values and indexed mean values..
  Minimum and maximum scores depend on the number of items in each domain which ranges from 3-7 items. A minimum score for a domain of 0 (worse) to a maximum of 15 for example and higher numbers are better.
Heart Rate | Baseline, 4, 8 and 12 weeks
  Heart rate data will be measured and compared from pre to post intervention
Heart rate variability data | Baseline, 4, 8 and 12 weeks
  Heart rate variability data collected for spectral analysis (vagal tone)
  Time domain analysis of vagal tone:
  Root mean squared of successive R-R interval difference change score between baseline and intervention time frames
  Frequency analysis of vagal tone:
  High frequency heart rate variability
Brief Fear of Movement scale adapted from the Tampa Scale of Kinesiophobia 11 (TSK-11) | Baseline, 4, 8 and 12 weeks
  Self report scale of fear avoidance and somatic focus with 11 questions and responses ranging from Strongly disagree (1) to strongly agree (4) on a 4 point Likert Scale. Scores range from a minimum of 11 to a maximum of 44 points with higher scores indicating greater fear of pain, movement, and injury
Stanford Brief Activity Survey | Baseline, 4, 8 and 12 weeks
  2 question- self report of usual daily work and leisure time activity and activity intensity to classify 5 activity levels, ranging from inactive to very hard intensity, using established metabolic equivalents for activity levels.
  The first item describes 5 different patterns of on-the-job activity, ranging from mostly sedentary to hard physical labor (such as carrying heavy loads). Similarly, the second item describes 5 patterns of leisure-time activity, ranging from sedentary to regular vigorous activity, such as running, on 5 or more days per week. Respondents select the 1 pattern that best describes their on-the-job activity and the 1 pattern that best describes their leisure-time activity. Each response pattern includes a global statement about the activity and the dimensions of frequency, intensity, time, and type of activity
Western Ontario and McMaster Universities Osteoarthritis Severity Index (WOMAC- Stiffness scale | Baseline, 4, 8 and 12 weeks
  2 Likert Scale questions of self-report joint stiffness The test questions are scored on a scale of 0-4, which correspond to: none (0), mild (1), moderate (2), severe (3), and extreme (4).
  The minimum score is 0 and the maximum is 8 and larger scores indicate worse stiffness.
Customized Technology Adoption Survey | 12th Week
  Modified Technology adoption survey of phone app use.(12 -6 point Likert Scaled questions ranging from 0 Very strongly disagree to very strongly agree ) with larger scores indicating better ease of use, attitude towards use and intent to use. The minimum score is 0 and the maximum score is 72.
Post-Intervention Qualitative Interview | Between 8th and 12th Week
  Semi-structured qualitative interview regarding phone app usability (ease of use), acceptability (satisfaction), pain, fear of pain, physical activity,

CONTACTS AND LOCATIONS:
Overall Officials: Linda Larkey, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States